CLINICAL TRIAL: NCT05152550
Title: Factors Predicting Transformation of Non-severe Pre-eclampsia Into Pre-eclampsia With Severe Features
Brief Title: Factors Predicting Transformation of Non Severe Pre-eclampsia Into Pre-eclampsia With Severe Features
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahmed Nagy Abdul-Rahman Younis (Other)
Responsible Party: Sponsor-Investigator, Ahmed Nagy Abdul-Rahman Younis, Professor, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Other Study IDs: 122016
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group A: Cases diagnosed as Non-severe pre-eclampsia after exclusion of severity features
  Interventions: Other: Non-severe pre-eclampsia

INTERVENTIONS:
Other: Non-severe pre-eclampsia — Cases diagnosed as Non-severe pre-eclampsia after exclusion of severity features.

SUMMARY:
Preeclampsia is a multi-system progressive disorder characterized by the new onset of hypertension and proteinuria, or hypertension and significant end-organ dysfunction with or without proteinuria, in the last half of pregnancy or postpartum. The genesis of the disease is laid down in early pregnancy and is characterized anatomically by abnormal remodeling of the maternal spiral arteries at the placental site.

DETAILED DESCRIPTION:
Eclampsia was firstly reported in 2200 BC in papyri of ancient Egypt. Eclampsia is originally a Greek word ´eklampsis and means "bright light". For 2000 years, eclampsia was known as a disease of convulsions in late gestation that resolves by childbirth. Scientists of late 19th century recognized the similarity in the swollen appearance of pregnant women who had seizures and explained all by the onset of glomerulonephritis with proteinuria. With the advanced noninvasive blood pressure measurement, it was observed that those women had increased blood pressure and not a long time before understanding that proteinuria and arterial hypertension occurrence before seizures. Thus, it was defined as "pre-eclampsia" that now it is a life-threatening condition for both the mother and the fetus.

Nowadays, hypertensive disorders during pregnancy, with an incidence that varies according to different measures, can exceed 10% in some population. Between multiple causes of maternal mortality and morbidity Pre-eclampsia and eclampsia are the second or third. [2]

A study made by WHO between 2003 and 2009 ranked hypertensive disorders as a cause of maternal deaths in the second grade, occurring in 14% of the cases, and in the first grade was hemorrhagic causes, responsible for 27.1%. [3] The 20th week of gestation is a period of interest as it is the landmark in the classification of hypertensive disorders because it is the time of the second wave of chorionic invasion. Thus hypertensive disorders were classified into two groups. The first one is before 20 weeks of gestation and includes essential chronic or secondary hypertension, white coat hypertension, "Masked" hypertension. The second group which appears at or after 20 weeks of gestation includes transient gestational hypertension, gestational hypertension, and pre-eclampsia.

In 2013, the American College of Obstetricians and Gynecologists (ACOG) replaced the term "severe pre-eclampsia" with the term "preeclampsia with severe features" which means systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥110 mmHg on at least 2 occasions, at least 4 hours apart after 20 weeks of gestation in a previously normotensive patient (with or without proteinuria) and the new onset of 1 or more of the following features:

A. Symptoms: Epigastric pain, hypochondrial pain, Cerebral or visual symptoms (e.g., new-onset and persistent headaches not accounted for by alternative diagnoses and not responding to usual doses of analgesics, blurred vision, flashing lights or sparks, scotomata).

B. Signs: Pulmonary edema and/or generalized edema.

C. Laboratory findings:

* Proteinuria ≥ 0.3 gm in a 24-hour urine specimen or protein/creatinine ratio ≥ 0.3 (mg/mg) (30 mg/m.mol) in a random urine specimen or dipstick ≥2+ if a quantitative measurement is unavailable.
* Platelet count <100,000/µL.
* Serum creatinine >1.1 mg/d L (97.2 µmol/L) or doubling of the creatinine concentration in the absence of another renal disease.
* Liver transaminases are at least twice the upper limit of the normal concentrations for the local laboratory.

In contrast to older criteria, the 2013 criteria severity features do not include proteinuria >5 g/24 hours and fetal growth restriction as features of severe disease.

So non-severe pre-eclampsia means that systolic BP from 130 to less than 160 mmHg, diastolic BP from 80 to less than 110 mmHg, and Proteinuria ≥ 0.3 gm in a 24-hour urine specimen or protein/creatinine ratio ≥ 0.3 (mg/mg) (30 mg/m.mol) in a random urine specimen or dipstick ≥2+ if a quantitative measurement is unavailable without the presence of the above-mentioned severity features.

In a woman with chronic/preexisting hypertension, criteria for superimposed preeclampsia are the new onset of proteinuria, significant end-organ dysfunction, or both after 20 weeks of gestation. For women with chronic/preexisting hypertension who have proteinuria prior to or in early pregnancy, superimposed preeclampsia is defined by worsening or resistant hypertension (especially acutely) in the last half of pregnancy or development of signs or symptoms of the severe end of the disease spectrum.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age above 20 weeks of gestation.
2. Cases diagnosed as Non-severe pre-eclampsia after exclusion of severity features which include:

   * Systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥110 mmHg.
   * Symptoms of central nervous system dysfunction of new onset such as Photopsia, scotomata, cortical blindness, retinal vasospasm, and severe headache.
   * Hepatic abnormality: Severe persistent right upper quadrant or Epigastric pain or serum transaminase concentration ≥2 times the upper limit of the normal range, or both.
   * Thrombocytopenia: < 100,000 platelets/µL.
   * Pulmonary edema.

Exclusion Criteria:

1. Vesicular mole (complete or incomplete).
2. Any cause of Albuminuria rather than PET such as (chronic kidney disease, type1 Diabetes mellitus.)
3. Any liver disease (Acute liver diseases cause increased liver transaminases and chronic liver diseases cause decreased production of albumin and transaminases.)
4. Any autoimmune disease that affects blood vessels or PLT count such as (ITP, TTP, SLE and rheumatoid arthritis.)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cases diagnosed as Non-severe pre-eclampsia after exclusion of severity features
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
severe pre-eclampsia | 4 months
  predicting transformation of non-severe pre-eclampsia in to pre-eclampsia with severe features

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Samy, MD, Principal Investigator — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No